CLINICAL TRIAL: NCT06360185
Title: Retrospective Study Investigating the Clinical Characteristic of Patients with Acute Presentation for Asthma to the A+E Department in a Busy Acute Hospital in England UK in Era of Biological Therapy for Asthma Between Jan 2019 & Jan 2024
Brief Title: Retrospective Study of Patients with Acute Presentation for Asthma to an Emergency Department in UK (RAPAE)
Acronym: RAPAE
Status: Not yet recruiting | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Asthma V2 October 2023
Record Dates: First submitted 2023-12-15; First posted 2024-04-11 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-03

CONDITIONS: Asthma Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Asthmatics presenting to the emergency department in NNUH over 5 years: Asthmatics presenting to the emergency department in NNUH over 5 years

SUMMARY:
Study team will obtain a list of all patients who have been seen in A+E over the past 6 years with a discharge diagnosis of asthma. Their history will be reviewed from their A+E notes. Team will obtain weight and height from Electronic prescribing tool and will obtain compliance information and past medical history from participant's GP records. Team will use participant's postcode to word out socio economic status quintile using office of national statistics tool. The following information will be taken from hospital documentation and from GP records.

DETAILED DESCRIPTION:
1. How many previous admissions in past one year (12 months)
2. How many presentations to A+E in previous one year (12 months)
3. Diagnosis not confirmed therefore not on any ICS
4. Poor compliance (less than 75% of ICS and/or LABA and/or LAMA and/or leukotriene prescriptions picked up in past year)
5. Recent presentation and maintenance therapy not increased (primary care or secondary care issue)
6. Is patient overweight BMI
7. Is patient on hormonal therapy, OCP, HRT, male hormones
8. Social class quintile from post code of address using ONS calculator
9. Ethnically diverse (see appendix)
10. First Eosinophil count on index admission
11. Highest eosinophil count in past (ever) and date
12. Treatment for diabetes type 2
13. Treatment for diabetes type 1
14. Treatment for hypertension
15. Smoker ever (pack year) when gave up__________

After obtaining this information study team will use simple statistical methods such as frequency and associations with confidence intervals to investigate which factors are associated with frequency of presentation to A+E. They will ascertain the frequency of patients who are on maximum therapy and may benefit from biological therapy, especially if they have raised eosinophils in the past year.

ELIGIBILITY:
Inclusion Criteria:

* All Asthmatics patients who attend Emergency department over 5 years

Exclusion Criteria:

* None Asthmatics.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The gender split changes with age: at age 11 years the relative risk of boys compared to girls within asthma population is 1.1 and by age 16 years the relative risk is 0.669. This change in gender association for asthma is poorly understood but highlights the complexities of asthma epidemiology. Adult asthma patients are more likely to be female and the study team would like to investigate if hormonal factors are related to reasons for presentation. This is difficult to elucidate in a retrospective study so the team is hoping that this study will inform them so they can undertake a prospective funded study regarding this service.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | 5 years
  Information will be taken from hospital documentation and from GP records.
Change in body height | 5 years
  Information will be taken from hospital documentation and from GP records.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiyah Hand, FRPC, Principal Investigator — Consultant Respiratory Physician

IPD SHARING:
Plan to Share IPD: Undecided